CLINICAL TRIAL: NCT00227942
Title: Understanding the Role That Hot Flashes and Sleep Disruption Play in the Effect of Estrogen Replacement Therapy on Mood in Perimenopausal and Postmenopausal Women
Brief Title: Estrogen for Treating Depression in Menopausal Women With Hot Flashes and Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadine Joffe, MD (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Hadine Joffe, MD, Director of Research at the Center for Women's Mental Health, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23MH066978 (NIH); K23MH066978 (NIH); DATR AK-TNAI1
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
Keywords: Women; Menopause; Depression; Hot flash; Insomnia; Sleep Disruption; Estrogen Replacement Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Hot Flashes | interventions — Estrogen Replacement Therapy; Estradiol; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive estrogen replacement therapy
  Interventions: Drug: Estrogen Replacement Therapy
- 2 (Experimental): Participants will receive treatment with zolpidem
  Interventions: Drug: Zolpidem
- 3 (Placebo Comparator): Participants will receive treatment with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Estrogen Replacement Therapy — 17-b-Estradiol Patch, .05 mg/day; applied for 7 days
  Other Names: Climara
  Arms: 1
Drug: Zolpidem — 10 mg/day, po qhs
  Other Names: Ambien
  Arms: 2
Drug: placebo — placebo
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of estrogen replacement therapy in treating depression in menopausal women with hot flashes and insomnia.

DETAILED DESCRIPTION:
Estrogen is a hormone that plays an important part in the development of the female reproductive system. During menopause, estrogen levels drop significantly. The drop in estrogen may cause physiologic and psychological changes in women; common symptoms include hot flashes, sweating, insomnia, and irritability. In addition, approximately 10% of menopausal women experience depression. Estrogen replacement therapy (ERT) is often prescribed to alleviate these symptoms. It is not known, however, exactly how ERT treats depression. It may indirectly decrease depression by alleviating insomnia associated with hot flashes, or it may directly improve mood and decrease depression by altering chemicals in the brain. The purpose of this study is to gain insight into how ERT treats depression and to develop strategies to reduce depression in menopausal women. In turn, these findings may help categorize populations of women whose depression should be treated with ERT versus nonhormonal therapies.

In this 9-week study, participants will be randomly assigned to receive ERT, a sleeping pill, or placebo. Study visits will occur at baseline and Weeks 2, 4, 6, and 9; at each study visit, blood pressure will be monitored, and standardized psychological tests and questionnaires will be used to assess the participant's level of depression and reported quality of life outcomes. Blood will be drawn at baseline and Week 9 to measure estrogen and follicle stimulating hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal or postmenopausal status
* Surgical menopause or hysterectomy with one or both ovaries preserved if serum follicle stimulating hormone is greater than 20 IU/L
* Diagnosed with mild to moderate clinical depression
* Currently experiencing moderate to severe hot flashes
* Currently experiencing insomnia caused by nocturnal hot flashes
* Normal mammogram within the 2 years prior to study entry
* Willing to use an effective form of contraception throughout the study if perimenopausal and sexually active

Exclusion Criteria:

* Current severe depression or history of severe depression within the 5 years prior to study entry
* Suicidal or homicidal ideation
* Psychotic symptoms
* History of any psychiatric disorder (e.g., psychosis, bipolar disorder, panic disorder, obsessive-compulsive disorder, or anorexia nervosa)
* History of any substance abuse (including alcohol abuse) within the 5 years prior to study entry
* Regular use of hormonal medications within the month prior to study entry
* Regular use of hypnotic drugs, antidepressants, or over-the-counter drugs known to influence hot flashes, sleep, or mood within the 2 weeks prior to study entry
* Intolerance to estrogen therapy or informed that estrogen therapy is medically inadvisable

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2003-08; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Improvement of mood; measured by the Montgomery-Asberg Depression Rating Scale | Measured at at baseline and Weeks 2, 4, 6, and 9

SECONDARY OUTCOMES:
Quality of life indicators; measured by the Quality of Life Inventory | Measured at at baseline and Weeks 2, 4, 6, and 9

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD, MSC, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Perinatal and Women's Mental Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Galvan T, Camuso J, Sullivan K, Kim S, White D, Redline S, Joffe H. Association of estradiol with sleep apnea in depressed perimenopausal and postmenopausal women: a preliminary study. Menopause. 2017 Jan;24(1):112-117. doi: 10.1097/GME.0000000000000737. PMID 27648659
- See also: Click here for the Massachusetts General Hospital Center for Women's Mental Health web site. — http://www.womensmentalhealth.org